CLINICAL TRIAL: NCT05576376
Title: Management of Intractable Plantar Fasciitis by Plantar Fascia Release Compared With Plantar Displacement Calcaneal Osteotomy: Randomized Control Study
Brief Title: Calcaneal Osteotomy for Intractable Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, El-Taher Alaa Eldin Ahmed Eid, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: plantar fasciitis
Record Dates: First submitted 2022-10-04; First posted 2022-10-12 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Plantar Fascitis
Keywords: intractable plantar fasciitis; heel spur; anteromedial heel pain
MeSH Terms: conditions — Heel Spur

STUDY DESIGN:
Intervention Model Description: We aim to achieve 35% percentage difference between both techniques with 80% power at a 5% (two-sided) significance level with alpha error 5%. For this power, a sample size of 54 patients will be required with assuming 10% drop out. So, a total of 60 patients will be enrolled (30 patients in each arm).
Who Masked: Outcomes Assessor
Masking Description: Each patient will be randomly assigned to his group using quick Calcs methodfor randomization (https://www.graphpad.com/quickcalcs/randomize1/) either group A (plantar fascia open release) or group B (Plantar fascia endoscopic release) or group C( calcaneal osteotomy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- plantar fascia release (Experimental): plantar fascia open release Longitudinal incision at the medial heel, Exposure of the plantar fascia at its origin on the medial plantar calcaneus. Medial incision of the plantar fascia preserving the lateral portion.. Exposure of the abductor hallucis muscle. Incision of the superficial fascia of the muscle. Retraction of the muscle belly und incision of the deep portion of the fascia, decompression of the first calcaneal branch of the lateral plantar nerve (Baxter's nerve) in cases of its being compressed.
  Postoperative management: Two weeks partial weight bearing. Progressively weight bearing using a shoe with a stiff sole for another 4 weeks.
  Interventions: Procedure: plantar fascia open release
- Plantar fascia endoscopic release (Experimental): We will draw a line distally from the posterior aspect of the medial malleolus to the intersection of the medial origin of the plantar fascia at the calcaneal tuberosity. A skin incision will be made, and medial portal will be performed at this location. Blunt dissection will be performed to clear the subcutaneous tissue from the plantar fascia with caution to avoid lesion of the calcaneal nerve medial branch.
  Interventions: Procedure: plantar fascia endoscopic release
- Clacaneal osteotomy (Experimental): calcaneal osteotomy skin incision will be oblique and directed from the inferoposterior edge of the lateral malleolus to the inferior edge of the calcaneal body, and subperiosteal exposure of the lateral calcaneal wall will be performed. Osteotomy will be performed from 1 cm anterior of the calcaneal attachment of the plantar fascia to 1 cm anterior of the calcaneal attachment of the Achilles tendon. After the osteotomy, approximately 5 mm plantar displacement of the proximal fragment, which include attachment of the plantar fascia, will be performed. Fixation after the osteotomy will be performed under an image intensifier using one cannulated cancellous screws 4.5 mm in diameter, which will be inserted from the infero-medial of the calcaneal tuberosity to the distal fragment
  Interventions: Procedure: calcaneal osteotomy for intractable plantar fasciitis

INTERVENTIONS:
Procedure: calcaneal osteotomy for intractable plantar fasciitis — plantar displacement calcaneal osteotomy
  Arms: Clacaneal osteotomy
Procedure: plantar fascia open release — open partial release with or without baxter's nerve decompression
  Arms: plantar fascia release
Procedure: plantar fascia endoscopic release — endoscopic partial plantar fascia release
  Arms: Plantar fascia endoscopic release

SUMMARY:
The aim of this study is to clarify the efficacy of plantar displacement calcaneal osteotomy for intractable plantar fasciitis by decreasing the tension of the plantar fascia around the calcaneal attachment while keeping the plantar fascia intact and comparing it with the plantar fascia release in pain control, job return and foot arch preservation.

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is the most common cause of heel pain accounting for 15% of all foot symptoms requiring medical care and 1% of patient visits to orthopaedic surgeons in the United states.

The diagnosis is straight forward; the challenge is finding an effective and economic first line treatment. The annual costs of plantar fasciitis are $284 million, that does not include opportunity cost from lost work and wages, societal burden, and psychologic burden.

Histologic examination shows myxoid degeneration with fragmentation and degeneration of the plantar fascia and supports being a degenerative fasciitis without inflammation. Therefore, plantar fasciopathy is a more accurate descriptor.

Treatment is largely nonoperative, with 85% to 90% of patients experiencing resolution of symptoms within 6-12 months. Partial or complete plantar fasciotomy, either open or endoscopic is indicated only for intractable cases with failed conservative treatment.

Fascia release, being the main surgery, sometimes accompanied by complications, one of which is lateral column pain due to loss of the longitudinal arch height caused by the release of the plantar fascia with no consensus regarding the amount of the plantar fascia which should be released in order to relieve pain without causing lateral column pain.

To avoid this complication, we need to study the efficacy of calcaneal osteotomy for the surgical treatment of PF. Does the calcaneal osteotomy is an effective alternative surgical treatment option compared to the standard plantar fascia release in cases of resistant PF?

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with age range from 18 to 65 years with unilateral or bilateral PF after clinical and radiological diagnosis confirmation, who had failed conservative treatment for at least 6 months or recurrent cases after steroid injection

Exclusion Criteria:

1. All other causes of heel pain including seronegative arthropathies, rheumatoid arthritis in bilateral cases, abscess or neoplasm affecting the soft tissue, and bone occult fracture or infection.
2. age groups below 18 years old and above 65 years old.
3. Plantar fasciitis cases with pes planus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
the change in the American Orthopaedic Foot and Ankle Society Ankle Hindfoot Scale (AOFAS score) | 6 months after surgery
  score of 100 points.higher score means better function with less pain and good alignment

IPD SHARING:
Plan to Share IPD: No